CLINICAL TRIAL: NCT02394704
Title: Graduated Sensory Salience as an Intervention for Intrusive Negative Thinking
Brief Title: Intervention for Intrusive Negative Thinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Liberos LLC (Industry)
Responsible Party: Principal Investigator, Greg Siegle, Associate Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PRO13040640
Record Dates: First submitted 2015-03-03; First posted 2015-03-20 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Intrusive Negative Thinking
Keywords: Rumination; Sensory processing; Non-pharmacological intervention; Depression; Anxiety; PTSD
MeSH Terms: conditions — Rumination Syndrome; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Graded sensory attention training (Experimental): Sensory stimuli will begin at a maximal tolerable intensity and decrease in intensity throughout the training, to shift from involuntary to voluntary attentional focus.
  Interventions: Other: Sensory attention training
- Non-graded sensory attention training (Active Comparator): Sensory stimuli will begin and be maintained at a minimal detectable intensity to maximize voluntary attentional training.
  Interventions: Other: Sensory attention training

INTERVENTIONS:
Other: Sensory attention training — Participants will be instructed to attend to sensory stimuli and to press a button as quickly and accurately as possible while ruminating. Stimuli will consist of vibration via a wearable subwoofer or non-painful electrical muscle stimulation (10Hz biphasic current with a pulse width of 200us with rectangular 2" electrodes placed on the back near the shoulders) or vibratory stimulation with a vibroacoustic element placed on the back near the shoulders. Up to four sessions will be approximately 45 minutes, over the course of two weeks.

SUMMARY:
Intrusive negative thinking styles such as rumination are typical of many psychiatric disorders, are difficult to treat, and predict poor treatment outcome. The investigators propose to evaluate a new intervention for negative thinking that capitalizes and builds on the preserved ability to attend to physical sensation. The investigators will examine changes in physiological mechanisms and symptoms.

DETAILED DESCRIPTION:
Intrusive negative cognitions are key features of many psychiatric disorders, are difficult to treat, and predict poor outcomes in conventional and neurobehavioral interventions. Here, we evaluate the extent to which a novel intervention capitalizing on a preserved neurocircuitry for attending to evolutionarily salient somatosensory stimuli can be used to train attentional mechanisms to override otherwise pre-potent negative cognitions. The initial period will involve open-label intervention refinement and mechanistic evaluation of mechanism; N=35 individuals with high levels of intrusive negative cognitions and dysphoria will be assessed pre/post intervention in the graded sensory training condition. Success will suggest a new intervention pathway for a traditionally treatment-resistant dimension of psychopathology. The second phase will be a randomized trial of 70 participants equally allocated to graded and non-graded training conditions.

ELIGIBILITY:
Inclusion Criteria for all participants:

* Signed study consent document
* Native English speakers (learned English before age 5)
* Right handed
* 20/30 vision or better
* Free from benzodiazepines and betablockers within 8 hours of evaluations

Subject specific Inclusion Criteria

* Endorsement of chronic and intrusive negative thinking
* High scores on rumination; Response Style Questionnaire (RSQ >= 44)
* Automatic Negative Thoughts Questionnaire (ATQ >= 48)
* Dysphoria; Quick Inventory of Depressive Symptomatology (QIDS>= 8)
* Must be in current treatment (either Intensive Outpatient Therapy, regular therapy sessions with a licensed provider, or close care by a psychiatrist). This is to ensure the research team is not the patient's only care provider, as this intervention is intended to be adjunct with therapy.

Exclusion Criteria:

* Refusal or inability to provide informed consent
* Current alcohol or substance dependence
* Psychotic disorders or psychosis
* Neurological disorders (stroke, Alzheimer's, Parkinson's, epilepsy, etc.)
* Inability to complete questionnaires in English. The justification is that many of the primary analyses involve assessment of change in self-reported symptoms using measures normed in English. Participants must thus be able to read those measures to give valid indications of the extent to which they have responded to the intervention.
* Current use of any psychotropic drugs thought to affect learning, including antipsychotics, anticonvulsants, stimulants, and anti-Parkinsonian drugs. Current is defined as within 2 weeks of testing, 4 weeks for fluoxetine.
* Chronic pain that could be exacerbated by transcutaneous electrical stimulation
* Having any eye problems or difficulties in corrected vision or hearing
* Having a North American Adult Reading Test (NAART) equivalent Full Scale Intelligence Quotient < 85
* Being pregnant. Determined by self-report at the interview and by a pregnancy test
* Severe or poorly controlled concurrent medical disorders that may cause thinking disruptions or require medication that could cause negative thinking
* Current use of medications that could cause affect thinking symptoms. That is, participants need to be able to think clearly to complete the proposed information processing tasks. And they need to be able to learn to be able to make use of the intervention. Medications which compromise clear thinking or which block learning will thus be considered exclusion criteria.
* Any implanted electrical device (pacemaker, vagus nerve stimulator implant, etc.) or prior treatment with a vagus nerve stimulator
* Underwent electroconvulsive therapy (ECT) < 9 months prior to study entry.
* People who have foreign objects in their body that are not cleared for safety at 3 Tesla scanning, such as aneurysm clips or pacemakers, will be excluded from the fMRI portion of the study.
* Participants deemed "not a good fit" for the study for other reasons (such as, but not limited to, continually arriving late or rescheduling, not being a trustworthy historian or accurate reporter of symptoms, being belligerent with study staff, or presenting an active suicide risk) can also be excluded.
* Any heart condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Sustained attention composite (computer based tasks and physiological measures) | two weeks (five intervention days)
  Sustained attention is operationalized by performance on computer-based tasks (sensitivity, reaction times) and associated physiological measures (pupil dilation, eye movements, heart rate, EEG) and central measures (fMRI derived reactivity in affect, somatosensory, and attention networks). These metrics will be interpreted together as a meta-analytic composite by counting the number of component measures with significant change in association with the intervention in comparison to a permutation-test derived critical number of indices change under the null hypothesis given the autocorrelation of the administered measures.

SECONDARY OUTCOMES:
Depressive severity (patient self-report) | two weeks (five intervention days)
  Clinical variables determined by patient self-report.
Rumination (patient self-report) | two weeks (five intervention days)
  Clinical variables determined by patient self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Greg J Siegle, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Oxford Building, Pittsburgh, Pennsylvania, United States